CLINICAL TRIAL: NCT03143842
Title: Can we Accelerate Learning in Tinnitus Participants Enrolled in the Vagus Nerve Stimulation (VNS) Study NCT01962558 /13-79?
Brief Title: Investigating Accelerated Learning in Tinnitus Participants Implanted With Vagus Nerve Stimulation
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Not enough participants
Sponsor: The University of Texas at Dallas (Other)
Collaborators: Defense Advanced Research Projects Agency (U.S. Federal Agency)
Responsible Party: Principal Investigator, Sven Vanneste, Associate professor, The University of Texas at Dallas
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 17-47
Record Dates: First submitted 2017-05-04; First posted 2017-05-08 (Actual); Last update posted 2022-01-28 (Actual); Status verified 2022-01

CONDITIONS: VNS Implanted Tinnitus Patients
Keywords: VNS; accelerate learning; memory
MeSH Terms: interventions — Vagus Nerve Stimulation

STUDY DESIGN:
Intervention Model Description: Within-subject design:
  To investigate whether VNS can accelerate learning and improve associative memory when learning word pairs, we will investigate the performance of VNS implanted participants on a Verbal Paired-Associate memory task and compare their performance on the words that were learned while paired with VNS in contrast to their performance on the words that were learned while unpaired with VNS and in contrast to their performance on the words that were learned without VNS (i.e. 3 types/groups of words: paired with VNS, unpaired with VNS and without VNS) during the first visit and 1 day,1 week and 1 month after their first visit.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Vagus Nerve Stimulation (Other): VNS paired with word pairs, VNS unpaired with word pairs, no VNS
  Interventions: Device: Vagus Nerve Stimulation

INTERVENTIONS:
Device: Vagus Nerve Stimulation — Delivering electrical pulses to the Vagus Nerve

SUMMARY:
The purpose of this study is to investigate whether it is possible to accelerate learning and improve memory performance in VNS implanted tinnitus participants by pairing VNS with a verbal paired-associate learning task.

DETAILED DESCRIPTION:
Associative memory refers to remembering the association between two items, such as a face and a name or a word in English and the same word in another language. It is not only important for learning, but it is also one of the first aspects of memory performance that is impacted by aging and by Alzheimer׳s disease. For decades, neuroscientists have investigated associative learning and memory and ways to accelerate and enhance associative learning and memory.

Vagus Nerve Stimulation (VNS) has been delivered to patient populations (e.g. depression, epilepsy, …) for more than 25 years and there has been some indications that this technique has effects on cognition, more specifically memory. Studies have investigated VNS as a way to improve memory performance and it has been shown in some studies to enhance memory in rats and humans. It has also demonstrated to produce changes in the electrophysiological and metabolic profile of forebrain and brainstem structures involved in learning and memory.

To investigate whether VNS can accelerate learning and improve associative memory when learning word pairs, we will investigate the performance of VNS implanted participants on a Verbal Paired-Associate memory task and compare their performance on the words that were learned while paired with VNS in contrast to their performance on the words that were learned while unpaired with VNS and in contrast to their performance on the words that were learned without VNS (i.e. 3 types/groups of words: paired with VNS, unpaired with VNS and without VNS) during the first visit and 1 day,1 week and 1 month after their first visit.

ELIGIBILITY:
Inclusion Criteria:

* 18-70 years old
* Native English speaker

Exclusion Criteria:

* Acquainted with the foreign language used in the learning task

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2017-04-27 (Actual); Primary Completion 2020-04-22 (Actual); Study Completion 2022-01-25 (Actual)

PRIMARY OUTCOMES:
Associative Memory assessed by a Verbal Paired-Associate test | Baseline session and 1 day, 1 week and 1 month after the baseline session
  Changes in performance in the Verbal Paired-Associate memory task is compared between three groups of learned word pairs (1) learned word pairs paired with VNS, (2) learned word pairs unpaired with VNS, (3) learned word pairs paired without VNS

CONTACTS AND LOCATIONS:
Overall Officials: Sven Vanneste, Ph.D., Principal Investigator — The University of Texas at Dallas
Locations (1):
- The University of Texas of Dallas, Richardson, Texas, United States

IPD SHARING:
Plan to Share IPD: Undecided